CLINICAL TRIAL: NCT00321971
Title: Prevention of Psychiatric Morbidity in AD Caregivers
Brief Title: Prevention of Depression in Spouses of People With Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Linda Garand, Associate Professor, Duquesne University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: K23MH070719 (NIH); K23MH070719 (NIH)
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Results first posted 2018-03-07 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Depression
Keywords: Anxiety; Mild Cognitive Impairment; MCI; Cognitive Impairment; Alzheimer's Disease; Caregiver Burden; Caregiver Stress; Family Dementia Caregiving; Spousal Dementia Caregiving
MeSH Terms: conditions — Depression; Anxiety Disorders; Cognitive Dysfunction; Alzheimer Disease; Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PST-MCI/AD Caregiving (Experimental): The experimental Intervention (PST-MCI/AD Caregiving) focuses on training in adaptive problem-solving attitudes and skills (Problem-Solving Therapy or PST). It was adapted from a manualized protocol for PST use in primary care. Our adaptation sought to enhance problem-solving skill levels of family caregivers as they began to face a variety of potential caregiving stressor.
  Interventions: Behavioral: PST-MCI/AD Caregiving
- NT-MCI/AD Caregiving (Active Comparator): The comparison Intervention (Caregiver Nutritional Training (NT-MCI/AD) was based on the United States Department of Health and Human Services (USDHHS) "2005 My Pyramid Dietary Guidelines for Americans over Age 50." We chose a nutrition-based comparison intervention because information about dietary practices is not likely to affect mental health outcomes. The NT intervention was matched to the PST-based intervention in terms of number and duration of sessions.
  Interventions: Behavioral: NT-MCI/AD Caregiving

INTERVENTIONS:
Behavioral: PST-MCI/AD Caregiving — The PST-based intervention will train participants to effectively use problem-solving skills with the aim of strengthening their ability to cope and preventing the onset or worsening of depressive and anxiety disorders. Participants received 2 phases of treatment; the first phase involved 6 sessions conducted in the caregiver's home approximately 2 weeks apart, each lasting approximately 1.5 hours. The second phase included three telephone contacts (approximately 2 weeks apart) to reinforce principles taught during the first phase, each lasting approximately 45 minutes.
  Arms: PST-MCI/AD Caregiving
Behavioral: NT-MCI/AD Caregiving — The nutritional education program will be based on the new USSDA dietary recommendations. Participants received 2 phases of treatment; the first phase involved 6 sessions conducted in the caregiver's home approximately 2 weeks apart, each lasting approximately 1.5 hours. The second phase included three telephone contacts (approximately 2 weeks apart) to reinforce principles taught during the first phase, each lasting approximately 45 minutes.
  Arms: NT-MCI/AD Caregiving

SUMMARY:
This study evaluates the effectiveness of a problem-solving training program in preventing depression in the spouses or family caregivers of persons with mild cognitive impairment or early dementia.

DETAILED DESCRIPTION:
People with a diagnosis of mild cognitive impairment (MCI) have an estimated 12% probability each year of progressing to a dementing disorder. Pilot data suggest that the spouses of people with MCI begin to adopt the caregiver role and its burdens as they cope with this condition. Although levels of caregiver burden and psychiatric illness are lower than those typically observed in family dementia caregiving samples, our findings suggest that MCI spousal caregivers have already begun to experience distress associated with elevated caregiver burden. In order to protect the mental health and well-being of caregivers as they cope with their spouses' current and future health care needs, it may be ideal to implement selective preventive strategies while they are in the very earliest stages of caregiving. This study evaluates the effectiveness of a problem-solving training program in preventing depression in the spouses or significant others of people with MCI.

Participants in this open-label study are randomly assigned to receive either a self-management intervention targeted at problem-solving training or an attention-matched intervention targeted at nutritional education. The self-management intervention trains participants to effectively use problem-solving skills with the aim of strengthening their ability to cope with burdens of caregiving and preventing the onset or worsening of depression. The nutritional education program is based on the new United States Department of Health and Human Services 2005 dietary recommendations. All participants attend weekly individual training sessions, either in their home or another convenient location for a total of 6 weeks. At the end of 6 weeks, participants receive a weekly phone call for an additional 3 weeks to support the training they received. Follow-up data is collected at Months 1, 3, 6, and 12 post-intervention. If a participant's spouse is diagnosed with dementia during the study, additional follow-up data is collected after the Month 12 visit.

ELIGIBILITY:
Inclusion Criteria:

* Spouse or non-married partner of a patient being treated at the University of Pittsburgh Alzheimer's Disease Research Center (ADRC) for a new or subsequent diagnosis of MCI

Exclusion Criteria:

* Does not speak English
* Cohabitating adult child of a person with MCI
* Resides in an institutional or assisted-living setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2007-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda J. Garand, PhD, Principal Investigator — The University of Pittsburgh School of Nursing
Locations (2):
- United States (2):
  - University of Pittsburgh Alzheimer's Disease Research Center (ADRC), Pittsburgh, Pennsylvania
  - Duquesne Univeristy, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garand L, Dew MA, Eazor LR, DeKosky ST, Reynolds CF 3rd. Caregiving burden and psychiatric morbidity in spouses of persons with mild cognitive impairment. Int J Geriatr Psychiatry. 2005 Jun;20(6):512-22. doi: 10.1002/gps.1318. PMID 15920711
- [Result] Garand L, Rinaldo DE, Alberth MM, Delany J, Beasock SL, Lopez OL, Reynolds CF 3rd, Dew MA. Effects of problem solving therapy on mental health outcomes in family caregivers of persons with a new diagnosis of mild cognitive impairment or early dementia: a randomized controlled trial. Am J Geriatr Psychiatry. 2014 Aug;22(8):771-81. doi: 10.1016/j.jagp.2013.07.007. Epub 2013 Oct 8. PMID 24119856
- [Derived] Garand L, Morse JQ, ChiaRebecca L, Barnes J, Dadebo V, Lopez OL, Dew MA. Problem-solving therapy reduces subjective burden levels in caregivers of family members with mild cognitive impairment or early-stage dementia: Secondary analysis of a randomized clinical trial. Int J Geriatr Psychiatry. 2019 Jul;34(7):957-965. doi: 10.1002/gps.5095. Epub 2019 Apr 17. PMID 30868641

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The University of Pittsburgh ADRC patient registry was searched for all cases diagnosed with MCI in the 6 months before the start of data collection and new cases of MCI or early dementia (any type) diagnosed at the ADRC during the subsequent 46-month time frame. Participants had to live with the person with MCI or early dementia
Groups:
- PST-AD/MCI Caregiving: The experimental Intervention focuses on training in adaptive problem-solving attitudes and skills (Problem-Solving Therapy or PST). It sought to enhance problem-solving skill levels of family caregivers as they began to face a variety of potential caregiving stressors. During the first session, participants received written and verbal education about the family caregiving role, the link between problems, overwhelming stress, symptoms of depression or anxiety, and the rationale for problem-solving training. In subsequent sessions, participants received written instructions and coaching in the systematic application of PST. Participants were asked to keep a record of their problem-solving efforts between sessions and questions they had related to the application of PST. These records were used as a basis for discussion during both phases of the intervention.
- NT-MCI/AD Caregiving: The comparison Intervention (Nutritional Training (NT-MCI/AD caregiving) was based on the United States Department of Health and Human Services (USDHHS) "2005 My Pyramid Dietary Guidelines for Americans over Age 50." We chose a nutrition-based comparison intervention because information about dietary practices is not likely to affect mental health outcomes. The NT intervention was matched to the PST-based intervention in terms of number and duration of sessions.
Period: Overall Study
Arm/Group | PST-AD/MCI Caregiving | NT-MCI/AD Caregiving
Started | 36 (Subject recruitment began in February 2007 and ended in December 2011) | 37
Completed | 28 | 26
Not Completed | 8 | 11

BASELINE CHARACTERISTICS:
Population: Of the 73 subjects enrolled in the study, 54 (71%) completed the study. Using an intention-to- treat approach, we performed a repeated-measures linear mixed effects analysis with the total sample (N=73) .
Groups:
- Problem Solving Training (PST): The experimental Intervention focuses on training in adaptive problem-solving attitudes and skills (Problem-Solving Therapy or PST). It sought to enhance problem-solving skill levels of family caregivers as they began to face a variety of potential caregiving stressors. During the first session, participants received written and verbal education about the family caregiving role, the link between problems, overwhelming stress, symptoms of depression or anxiety, and the rationale for problem-solving training. In subsequent sessions, participants received written instructions and coaching in the systematic application of PST. Participants were asked to keep a record of their problem-solving efforts between sessions and questions they had related to the application of PST. These records were used as a basis for discussion during both phases of the intervention.
- Nutritional Training (NT): The comparison Intervention (Nutritional Training (NT-MCI/AD caregiving) was based on the United States Department of Health and Human Services (USDHHS) "2005 My Pyramid Dietary Guidelines for Americans over Age 50." We chose a nutrition-based comparison intervention because information about dietary practices is not likely to affect mental health outcomes. The NT intervention was matched to the PST-based intervention in terms of number and duration of sessions. Participants were asked to keep a record of menu planning, eating habits between session, and any questions they had related to the application of NT. These records were used as a basis for discussion during both phases of the intervention
- Total: Total of all reporting groups
Arm/Group | Problem Solving Training (PST) | Nutritional Training (NT) | Total
Number analyzed (Participants) | 36 | 37 | 73
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.4 (8.0) | 63.4 (13.7) | 64.98 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 36 | 37 | 73
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 35 | 37 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 37 | 73

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptoms
Description: Depressive symptoms were measured with Center for Epidemiological Studies - Depression Scale (CES-D). The CES-D was designed as a self-report measure of depressive symptoms in nonpsychiatric subjects and has been used with spousal dementia caregiving populations with no report of negative psychological effects. It is composed of 20 items, each rated on a 4-point response scale corresponding to the frequency of the symptom in the preceding week. The possible range of CES-D scores is 0-60, with a higher score indicating more severe symptoms. A cutoff score of 16 or greater is indicative of individuals at high risk for clinical depression. The CES-D was chosen because of its relatively high internal reliability (Cronbach's alpha = .88) and predictive validity for the diagnosis of depression.
Time Frame: Baseline and 1-, 3-, 6-, and 12- months post-treatment
Population: Using an intention-to-treat approach, we performed a repeated-measures linear mixed effects analysis for each study outcome. This analysis included group assignment (PST-MCI/AD Caregiving vs NT), type of caregiver (MCI versus dementia), and time (baseline, 1-, 3-, 6-, and 12-month follow-up). The depression data were log-transformed for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Problem Solving Intervention: The experimental Intervention (PST-MCI/AD Caregiving) focuses on training in adaptive problem-solving attitudes and skills (Problem-Solving Therapy or PST). It was adapted from the work of Areán and colleagues, who developed a manualized protocol for PST use in primary care. Our adaptation sought to enhance problem-solving skill levels of family caregivers as they began to face a variety of potential caregiving stressor.
  Problem-solving therapy: The self-management intervention will train participants to effectively use problem-solving skills with the aim of strengthening their ability to cope and preventing the onset or worsening of depressive and anxiety disorders. All participants attend weekly individual training sessions, either in their home, another convenient location, or by telephone for a total of 9 weeks.
- Nutritional Intervention: The comparison Intervention (Caregiver Nutritional Training (NT-MCI/AD) was based on the United States Department of Health and Human Services (USDHHS) "2005 My Pyramid Dietary Guidelines for Americans over Age 50." We chose a nutrition-based comparison intervention because information about dietary practices is not likely to affect mental health outcomes. The NT intervention was matched to the PST-based intervention in terms of number and duration of sessions.
  Nutritional education program: The nutritional education program will be based on the new USDA dietary recommendations. All participants attend weekly individual training sessions, either in their home or another convenient location for a total of 6 weeks.
Arm/Group | Problem Solving Intervention | Nutritional Intervention
Number analyzed (Participants) | 36 | 37
units on a scale
  Baseline | 9.736 (1.594) | 11.785 (1.515)
  1 Month Follow-up | 8.880 (1.777) | 12.300 (1.715)
  3 Month Follow-up | 8.766 (1.927) | 13.157 (1.848)
  6 Month Follow-up | 6.885 (1.689) | 13.831 (1.637)
  12 Month Follow-Up | 6.475 (1.619) | 14.143 (1.571)
Statistical Analysis 1: Comparison: Problem Solving Intervention; Hypothesis: The experimental intervention group will endorse lower mean levels of depressive symptoms during follow-up than the study group receiving the comparison intervention; Test type: Superiority; p < .05, Mixed Models Analysis; Intention-to-treat model; Mean Difference (Final Values) = 0.421, 95% CI 2-sided [0.208 to 0.657], Standard Error of Mean .110 — The CES-D data were log-transformed for analysis

ADVERSE EVENTS:
Time Frame: Baseline, 1, 3, 6 and 12 months post intervention
Groups:
- Experimental Intervention: The experimental Intervention (PST-MCI/AD Caregiving) focuses on training in adaptive problem-solving attitudes and skills (Problem-Solving Therapy or PST). Participants received 2 phases of treatment; the first phase involved 6 sessions conducted in the caregiver's home approximately 2 weeks apart, each lasting approximately 1.5 hours. The second phase included three telephone contacts (approximately 2 weeks apart) to reinforce principles taught during the first phase, each lasting approximately 45 minutes.
  During the first session, participants received written and verbal education about the structure of sessions, MCI or dementia and the family caregiving role, the link between problems, overwhelming stress, and symptoms of depression, the relationship between low mood and reduced pleasurable activities, and the rationale for problem-solving training. In subsequent sessions, participants received written instructions and coaching in the systematic application of PST.
- Comparison/Control Intervention: The comparison Intervention (Caregiver Nutritional Training (NT-MCI/AD) was based on the USDHHS "My Pyramid Dietary Guidelines for Americans over Age 50." The NT intervention was matched to the PST-based intervention in terms of number and duration of sessions.
  During the first session, participants received written and verbal education about the structure of the sessions, MCI or dementia, and an overview of USDA Dietary Guidelines. Participants also completed a questionnaire about their current eating practices and activity level. In subsequent training sessions, the interventionist provided education related to the major food categories, discretionary calories, and tips and resources for menu planning. Participants were asked to keep a record of menu planning, eating habits between session, and any questions they had related to the application of NT. These records were used as a basis for discussion during both phases of the intervention.
Arm/Group | Experimental Intervention | Comparison/Control Intervention
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/37
Other Adverse Events (participants affected / at risk) | 0/36 | 0/37

LIMITATIONS AND CAVEATS:
The relatively small size and racial composition of the sample was a limitation. The generalizability of our findings are reduced by our focus on family caregivers who reside with the individual with cognitive impairment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes